CLINICAL TRIAL: NCT01803087
Title: A SINGLE-DOSE, OPEN LABEL, RANDOMIZED, 3-WAY CROSSOVER, CLINICAL PHARMACOLOGY STUDY OF CHF 1535 100/6 pMDI (FIXED COMBINATION OF BECLOMETHASONE DIPROPIONATE 100 µg PLUS FORMOTEROL FUMARATE 6 µg) WITH OR WITHOUT SPACER DEVICE VERSUS THE FREE COMBINATION OF LICENSED BECLOMETHASONE pMDI AND FORMOTEROL pMDI IN ASTHMATIC ADOLESCENT PATIENTS AND ONE OPEN ARM FOR ADULT PATIENTS AS CONTROL GROUP TREATED WITH CHF 1535 100/6 pMDI.
Brief Title: Single-Dose Clinical Pharmacology Study in Asthmatic Adolescent and Adult Patients
Acronym: ADO pMDI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CCD-1104-PR-0062
Record Dates: First submitted 2012-10-04; First posted 2013-03-04 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Asthma
Keywords: adolescents; adults
MeSH Terms: conditions — Asthma | interventions — Foster Home Care; Beclomethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CHF 1535 100/6 pMDI (Foster®) TEST 1 (Active Comparator): Adolescents CHF 1535 100/6, 4 puffs (total dose: BDP 400 µg/FF 24 µg) pMDI
  Interventions: Drug: Test treatments CHF 1535 100/6 pMDI (Foster®) TEST1
- CHF 1535 100/6 pMDI (Foster®) AeroChamber Plus™ (TEST 2). (Active Comparator): CHF 1535 100/6 pMDI (Foster®) using AeroChamber Plus™ spacer device in adolescents (TEST 2)
  Interventions: Drug: CHF 1535 100/6 pMDI (Foster®) using AeroChamber Plus™ (TEST 2).
- (Qvar®: BDP 400 µg)+(Atimos®: formoterol 24 µg) (Active Comparator): BDP 100 µg pMDI, 4 puffs (Qvar®, total dose: BDP 400 µg) + formoterol fumarate 6 µg pMDI, 4 puffs (Atimos®, total dose: formoterol 24 µg)
  Interventions: Drug: BDP pMDI 100 µg (Qvar®) plus formoterol fumarate pMDI 6 µg (Atimos®) (REF)
- CHF 1535 100/6, 4 puffs (total dose: BDP 400 µg/FF 24 µg) pMDI (Active Comparator): Adults CHF 1535 100/6, 4 puffs (total dose: BDP 400 µg/FF 24 µg) pMDI
  Interventions: Drug: CHF 1535 100/6 pMDI (Foster®) (CTR)

INTERVENTIONS:
Drug: Test treatments CHF 1535 100/6 pMDI (Foster®) TEST1
  Arms: CHF 1535 100/6 pMDI (Foster®) TEST 1
Drug: CHF 1535 100/6 pMDI (Foster®) using AeroChamber Plus™ (TEST 2).
  Arms: CHF 1535 100/6 pMDI (Foster®) AeroChamber Plus™ (TEST 2).
Drug: BDP pMDI 100 µg (Qvar®) plus formoterol fumarate pMDI 6 µg (Atimos®) (REF)
  Other Names: Free combination of BDP pMDI 100 µg (Qvar®) plus formoterol fumarate pMDI 6 µg (Atimos®) in adolescents (REF)
  Arms: (Qvar®: BDP 400 µg)+(Atimos®: formoterol 24 µg)
Drug: CHF 1535 100/6 pMDI (Foster®) (CTR)
  Other Names: CHF 1535 100/6 pMDI (Foster®) in adults (CTR)
  Arms: CHF 1535 100/6, 4 puffs (total dose: BDP 400 µg/FF 24 µg) pMDI

SUMMARY:
This clinical pharmacology want to investigate the systemic availability of BDP/B17MP (active metabolite of BDP) and formoterol after single oral inhalation of CHF 1535 100/6 pMDI with and without spacer device (AeroChamber Plus™) and in comparison to a free combination of BDP pMDI plus formoterol pMDI licensed products; this will be additionally compared to the systemic exposure in adults without the spacer device.

DETAILED DESCRIPTION:
The proposed clinical pharmacology study is aimed to investigate the systemic availability of BDP/B17MP (active metabolite of BDP) and formoterol after single oral inhalation of CHF 1535 100/6 pMDI (to reach a total dose of BDP 400 µg and formoterol 24 µg) with and without spacer device (AeroChamber Plus™) and in comparison to a free combination of BDP pMDI plus formoterol pMDI licensed products (to reach the same total dose of BDP and formoterol) in adolescent asthmatic patients. The systemic exposure to BDP/B17MP and formoterol after inhalation of CHF 1535 pMDI in adolescents will be additionally compared to the systemic exposure in adults without the spacer device.

The chosen doses correspond to the maximum daily dose of the two components administered as fixed combination.

ELIGIBILITY:
- Inclusion criteria

Patients will be enrolled if they meet all of the following criteria:

1. Male and female adolescents, aged ≥ 12 and < 18 years at the time of Screening Visit or male and female adults, aged ≥ 18 and ≤ 65 years at the time of Screening Visit.
2. Written informed consent obtained by the patient in case of adult patients and by parents/legal representative and by the minor (according to local regulation).
3. A diagnosis of asthma as defined in the GINA guidelines (updated 2010) 6 months before the screening visit.
4. Male/female adolescent and adult patients with asthma stable enough, according to GINA guidelines (updated 2010) and based on the Investigator's opinion, to allow a wash out period from inhaled BDP of 2 days before each single day study treatments and any ICS other than BDP of 1 day before each single day study treatments.
5. Male/female adolescents and adults asthmatic patients already treated with ICS or ICS/long-acting inhaled β2-agonists or using short-acting inhaled β2-agonists as reliever to control asthma symptoms.
6. Adolescents and adults with a forced expiratory volume in one second (FEV1) > 70% of predicted values (% pred) after withholding short acting β2-agonist treatment for a minimum of 6 h prior to screening or 24 hours in case of long acting β2-agonist.
7. Non- or ex-smokers who smoked less than 5 pack-years (e.g. < 20 cigarettes per day for 5 years) and stopped smoking for at least 1 year.
8. A cooperative attitude and ability to be trained about the proper use of pMDI with and without a spacer device and compliant to study procedures.
9. Body mass index (BMI) ≥18.5 and ≤ 32 kg/m2

   * Exclusion criteria

Patients will not be enrolled if one or more of the following criteria are present:

1. Pregnant or breast-feeding female patients. Sexually active female not using efficient contraception throughout the entire study period (e.g. oestro-progestatives, condoms, intrauterine devices). A urinary pregnancy test will be performed at screening and treatment visits (mandatory in the adult population and at discretion of the investigator in the adolescent population) in women of childbearing potential;
2. Having received an investigational drug within 2 months before the screening visit (Visit 1).
3. Diagnosis of COPD, in the adult patients, as defined by the current GOLD guidelines (updated 2010).
4. Known hypersensitivity to the active treatments.
5. Inability to perform the required breathing technique and blood sampling.
6. Hospitalization due to exacerbation of asthma within 1 month prior to the screening visit.
7. Lower respiratory tract infection within 1 month prior to screening visit.
8. Obesity, i.e. > 97% weight percentile by local standards.
9. Significant medical history of and/or treatments for cardiac, renal, neurological, hepatic, endocrine diseases, that may interfere with patient's safety, compliance, or study evaluations, according to the Investigator's opinion;
10. History of drug addiction or excessive use of alcohol (weekly intake in excess of 28 units alcohol; one unit being a glass of beer, wine or a measure of spirits), or excessive consumption of xanthine containing substances (daily intake in excess of 5 cups of coffee, tea, cola, etc) or psychological or other emotional problems likely to invalidate informed consent, or limit the ability of the subject to comply with the protocol requirements;
11. Treatment with a xanthine derivative (e.g. theophylline) formulations in the 4 weeks prior to screening;
12. Blood donation (450 mL or more) (for the adult population) or significant blood loss in the 12 weeks before the screening visit.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2012-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
AUC0-t of B17MP CHF 1535 100/6 pMDI with and without spacer vs free combination of BDP pMDI and formoterol pMDI | : pre-dose (within 5 min from dosing), 5 min; 15 min; 30 min; 1, 2, 4, 6 and 8 hr after inhalation.
  In adolescents, the systemic exposure of B17MP as AUC0-t, after inhalation of CHF 1535 100/6 pMDI with and without spacer device (AeroChamber Plus™) vs already licensed free combination of BDP pMDI and formoterol pMDI without spacer.

SECONDARY OUTCOMES:
AUC0-t, AUC0-inf, Cmax, tmax and t½ for BDP and formoterol | : pre-dose (within 5 min from dosing), 5 min; 15 min; 30 min; 1, 2, 4, 6 and 8 hr after inhalation.
  In adolescents, after inhalation of CHF1535 100/6 pMDI both with and without spacer vs a free combination of licensed BDP and Formoterol pMDIs.
AUC0-0.5h, AUC0-inf, Cmax, tmax and t½ for B17MP | : pre-dose (within 5 min from dosing), 5 min; 15 min; 30 min; 1, 2, 4, 6 and 8 hr after inhalation.
  In adolescents, after inhalation of CHF1535 100/6 pMDI both with and without spacer vs a free combination of licensed BDP and Formoterol pMDIs.
plasma glucose and plasma potassium AUC0-t; Cmin; Tmin; Cmax; Tmax | : pre-dose (within 5 min from dosing), 5 min; 15 min; 30 min; 1, 2, 4, 6 and 8 hr after inhalation.
  In adolescents, after inhalation of CHF 1535 100/6 pMDI with and without spacer (AeroChamber Plus™)vs fre combination
Heart rate as AUC0-8h of CHF 1535 100/6 pMDI | pre-dose (within 5 min from dosing), 5 min; 10 min; 15 min; 30 min; 1, 2, 4, 6 and 8 hr after inhalation.
  In adolescents, after inhalation of CHF1535 100/6 pMDI both with and without spacer vs free combination
FEV1; time everaged FEV1 value AUC0-8h; peak FEV1 | pre-dose; 30 min; 1, 2, 4, 6 and 8 hr after inhalation.
  In adolescents, after inhalation of CHF1535 100/6 pMDI both with and without spacer vs a free combination of licensed BDP and Formoterol pMDIs.

CONTACTS AND LOCATIONS:
Locations (1):
- Uniwersytecki Szpital Kliniczny nr 1, Lodz, Poland

REFERENCES:
- [Result] Kuna P, Govoni M, Lucci G, Scuri M, Acerbi D, Stelmach I. Pharmacokinetics and pharmacodynamics of an extrafine fixed pMDI combination of beclometasone dipropionate/formoterol fumarate in adolescent asthma. Br J Clin Pharmacol. 2015 Sep;80(3):569-80. doi: 10.1111/bcp.12640. Epub 2015 Jun 1. PMID 25808292
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=CCD-1104-PR-0062